CLINICAL TRIAL: NCT07398105
Title: A Clinical Study Comparing Virtual Reality and Mixed Reality Head-Mounted Displays for Dental Anxiety and Pain Control During Local Anesthesia in Children
Brief Title: Comparison of Virtual Reality and Mixed Reality Head-Mounted Displays for Dental Anxiety Control During Local Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Enes Mustafa AŞAR, Assistant professor, Selcuk University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBAE Thesis Project
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dental Anxiety
Keywords: Pediatric Dentistry; Virtual Reality; Mixed Reality; Dental Anxiety; Local Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Behavioral pain responses were assessed by two independent observers who were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) Group (Other): Children who preferred virtual reality distraction received audiovisual content through a head-mounted display during local anesthesia administration. The virtual reality mode provided a fully immersive environment intended to reduce dental anxiety and pain perception.
  Interventions: Behavioral: Audiovisual Distraction Using Head-Mounted Display
- Mixed Reality (MR) Group (Other): Children who preferred mixed reality distraction received audiovisual content through a head-mounted display during local anesthesia administration. The mixed reality mode allowed interaction with virtual content while maintaining partial awareness of the clinical environment to support anxiety and pain control.
  Interventions: Behavioral: Audiovisual Distraction Using Head-Mounted Display

INTERVENTIONS:
Behavioral: Audiovisual Distraction Using Head-Mounted Display — Participants received audiovisual distraction through a head-mounted display during local anesthesia administration. The intervention was delivered in two modes based on participant preference: a virtual reality (VR) mode providing a fully immersive audiovisual environment, and a mixed reality (MR) mode allowing interaction with virtual content while maintaining partial awareness of the clinical environment.

SUMMARY:
Dental anxiety is a common problem in children and may negatively affect cooperation, pain perception, and treatment success during dental procedures. Distraction techniques are widely used to reduce anxiety during dental treatment. In recent years, virtual reality (VR) and mixed reality (MR) technologies have been introduced as innovative audiovisual distraction methods in pediatric dentistry.

The aim of this randomized clinical study is to compare the effects of virtual reality and mixed reality head-mounted displays on dental anxiety and pain perception in children during local anesthesia administration. A total of 142 systemically healthy children aged 6 to 12 years who required dental treatment under local anesthesia were included. Participants were randomly assigned to either a VR group or an MR group.

Dental anxiety and pain levels were assessed using validated scales before and during local anesthesia administration. Behavioral responses and physiological parameters were also recorded. The results of this study will help determine whether VR or MR provides superior anxiety control during pediatric dental procedures.

DETAILED DESCRIPTION:
Dental anxiety in children is associated with increased pain perception, behavioral problems, and reduced treatment compliance. Managing anxiety during dental procedures is therefore a critical component of pediatric dental care. Conventional behavior guidance techniques may not always be sufficient, particularly during invasive procedures such as local anesthesia administration.

This randomized, parallel-group clinical trial was conducted to compare the effects of virtual reality (VR) and mixed reality (MR) head-mounted displays on dental anxiety and pain perception in pediatric patients. The study included 142 systemically healthy children aged between 6 and 12 years who required dental treatment under local anesthesia. Only children with positive or definitely positive behavior according to the Frankl Behavior Rating Scale were included.

Participants were randomly allocated into two groups: a VR group and an MR group. During local anesthesia administration, children in the VR group were exposed to a fully immersive virtual environment, while children in the MR group interacted with virtual content while maintaining partial awareness of the clinical environment.

Dental anxiety was evaluated using the Children's Fear Survey Schedule-Dental Subscale, and pain perception was assessed using the Wong-Baker FACES Pain Rating Scale. Behavioral pain responses during local anesthesia were scored using the FLACC scale by two independent observers. Heart rate measurements were recorded as a physiological indicator of anxiety. Interobserver reliability for behavioral assessments was also evaluated.

The primary outcome of the study was the change in dental anxiety levels during local anesthesia administration. Secondary outcomes included pain perception, behavioral responses, and physiological changes. The findings of this study aim to provide evidence regarding the effectiveness of VR and MR technologies as distraction tools for anxiety management in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 and 12 years.
* Systemically healthy children.
* Children requiring dental treatment under local anesthesia.
* Positive or definitely positive behavior according to the Frankl Behavior Rating Scale.
* Written informed consent obtained from parents or legal guardians.

Exclusion Criteria:

* Presence of systemic disease or neurological disorders.
* Visual or auditory impairment that could interfere with the use of head-mounted displays.
* History of epilepsy, vertigo, or motion sickness related to audiovisual stimulation.
* Negative or definitely negative behavior according to the Frankl Behavior Rating Scale.
* Refusal to use virtual reality or mixed reality devices.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2024-05-04 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Dental Anxiety Level During Local Anesthesia | Immediately before and during local anesthesia administration
  Dental anxiety levels were assessed using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS). Anxiety scores were recorded before and during local anesthesia administration to evaluate changes associated with virtual reality and mixed reality distraction methods.

SECONDARY OUTCOMES:
Pain Perception During Local Anesthesia | During local anesthesia administration
  Pain perception was evaluated using the Wong-Baker FACES Pain Rating Scale during local anesthesia administration.
Behavioral Pain Response Assessed by FLACC Scale | During local anesthesia administration
  Behavioral pain responses during local anesthesia administration were assessed using the FLACC (Face, Legs, Activity, Cry, Consolability) scale by two independent observers.
Heart Rate Changes During Local Anesthesia | Immediately before, after and during local anesthesia administration
  Heart rate was measured as a physiological indicator of anxiety before and during local anesthesia administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No